CLINICAL TRIAL: NCT03961997
Title: PHASE 1, OPEN-LABEL, FIXED SEQUENCE, 2-PERIOD STUDY TO INVESTIGATE THE EFFECT OF MULTIPLE DOSES OF MODAFINIL ON THE PHARMACOKINETICS OF SINGLE DOSE LORLATINIB (PF-06463922) IN HEALTHY PARTICIPANTS
Brief Title: Effect of Multiple Doses of Modafinil on the Pharmacokinetics of Single Dose Lorlatinib in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: B7461026; 2019-001455-40 (EudraCT Number)
Record Dates: First submitted 2019-05-22; First posted 2019-05-23 (Actual); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Adult; Drug Interactions; Healthy Volunteers; Humans
Keywords: Cytochrome P-450 CYP3A Inhibitors/metabolism; Cytochrome P-450 CYP3A Inhibitors/adverse effects; Cytochrome P-450 CYP3A Inhibitors/pharmacokinetics; Cytochrome P-450 CYP3A Inhibitors/pharmacology; Modafinil/adverse effects; Modafinil/pharmacokinetics; Modafinil/pharmacology
MeSH Terms: interventions — lorlatinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Lorlatinib 50 mg (Other): Participants will receive a single dose of lorlatinib 50 mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 50 mg on Day 15 of Period 2.
  Interventions: Drug: Lorlatinib 50 mg
- Lorlatinib 75 mg (Other): Participants will receive a single dose of lorlatinib 75mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 75 mg on Day 15 of Period 2.
  Interventions: Drug: Lorlatinib 75 mg
- Lorlatinib 100 mg (Other): Participants will receive a single dose of lorlatinib 100 mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 100 mg on Day 15 of Period 2.
  Interventions: Drug: Lorlatinib 100 mg

INTERVENTIONS:
Drug: Lorlatinib 50 mg — Participants will receive a single dose of lorlatinib 50 mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 50 mg on Day 15 of Period 2.
  Arms: Lorlatinib 50 mg
Drug: Lorlatinib 75 mg — Participants will receive a single dose of lorlatinib 75 mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 75 mg on Day 15 of Period 2.
  Arms: Lorlatinib 75 mg
Drug: Lorlatinib 100 mg — Participants will receive a single dose of lorlatinib 100 mg in Period 1. Participants will receive modafinil 400 mg daily for 19 days, and a single dose of lorlatinib 100 mg on Day 15 of Period 2.
  Arms: Lorlatinib 100 mg

SUMMARY:
The primary purpose of the study is to characterize the safety profile of lorlatinib in the presence of a moderate CYP3A4/5 inducer, modafinil. In another drug-drug interaction study for lorlatinib coadministered with a strong CYP3A4/5 inducer, rifampin, all participants experienced increases in liver enzymes after receiving the combination of a single dose lorlatinib (100 mg) with rifampin (600 mg daily (QD)) after multiple doses of rifampin. The AST and ALT continued to increase over the next 24-48 hours, but recovered below the upper limit of normal for all participants upon discontinuation of rifampin.

We hypothesize the combination of lorlatinib with the moderate CYP3A inducer modafinil will not have a safety findings related to liver enzyme elevation similar to what occurred in the study with rifampin and lorlatinib.

DETAILED DESCRIPTION:
This will be a Phase 1 study in approximately 16 healthy participants employing administration of a single dose of lorlatinib in the fasted state alone, and with multiple doses of modafinil 400 mg once daily. This study will consist of up to 3 lorlatinib treatment groups: 50, 75, or 100 mg single doses of lorlatinib given alone and in combination with multiple doses of modafinil.

Each enrolled participant will receive lorlatinib 50, 75, or 100 mg alone in Period 1 and then lorlatinib 50, 75, or 100 mg in combination with multiple dose modafinil in Period 2 after a washout period of at least 19 days between lorlatinib doses in Periods 1 and 2. A single PK sample is taken prior to lorlatinib dosing in each period. Following administration of lorlatinib in each period, participants will undergo serial PK sampling.

There will be 4 cohorts. Cohorts 1 to 3 will include 2 participants each, while Cohort 4 will include 10 participants. Participants in Cohorts 1 to 4 will be sequentially enrolled such that participants in a new cohort can receive their lorlatinib Period 2 dose only after participants from the prior cohort are 72 hours past their lorlatinib Period 2 combination dose (with modafinil) with no safety concerns. In addition, Cohorts 1 to 3 will employ sentinel dosing such that the second participant in each cohort can receive their lorlatinib Period 2 dose only after the first participant from the same cohort is 72 hours past their lorlatinib and modafinil Period 2 combination dose with no safety concerns. Participants in Cohort 4 may be dosed in parallel, as sentinel dosing of lorlatinib 100 mg will have been completed in Cohort 3. The overall study design will be identical in all 4 cohorts, with the only difference being the dose of lorlatinib administered.

The decision to dose subsequent cohorts during Period 2 with lorlatinib will be made after reviewing the totality of the participants' clinical picture for safety by the investigator. Furthermore, participants in subsequent cohorts will not be dosed if the following liver function abnormalities are observed during the 72 hour time frame for safety evaluation after lorlatinib dosing in Period 2.

For enrollment of each successive cohort, the period of safety evaluation will be at least 72 hours after the Period 2 lorlatinib dosing in the previous cohort. During Period 2, safety laboratory assessments including urinalysis, hematology and chemistry will be performed once daily from Day 14 through Day 20. Only after the review of safety labs for at least 72 hours after lorlatinib+ modafinil dosing during Period 2 of the previous cohort, will participants in a new cohort receive lorlatinib in combination with modafinil in their Period 2. Additional safety laboratory assessments may be performed at any additional times at the discretion of the investigator. If safety events of concern are observed in Cohorts 1, 2, or 3 during Period 2, this study will be terminated.

ELIGIBILITY:
Inclusion Criteria:

* Male and female participants who are overtly healthy as determined by medical evaluation including medical history, physical examination, laboratory tests, and ECG.
* Adequate Renal Function, including:

Estimated creatinine clearance ≥90 mL/min as calculated using chronic kidney disease epidemiology collaboration equation (CKD EPI). In equivocal cases, a 24 hour urine collection test can be used to estimate the creatinine clearance more accurately.

- Adequate Liver Function, including: Total serum bilirubin within normal limits (WNL). Aspartate and Alanine aminotransferase (AST and ALT) WNL. Alkaline phosphatase WNL.

* Participants who are willing and able to comply with all scheduled visits, treatment plan, laboratory tests, lifestyle considerations, and other study procedures.
* Male participants of childbearing potential must agree to use a highly effective method of contraception from the first screen throughout the study and for 97 days after the last dose of assigned treatment if male participant. A participant is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.
* Body mass index (BMI) of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).
* Capable of giving signed informed consent as described in Appendix 1, which includes compliance with the requirements and restrictions listed in the informed consent document (ICD) and in this

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* History of human immunodeficiency virus (HIV) infection, hepatitis B, or hepatitis C; positive testing for HIV, hepatitis B surface antigen (HepBsAg), or hepatitis C antibody (HCVAb). A positive hepatitis B surface antibody (HepBsAb) serology indicating Hepatitis B vaccination is allowed.
* Other acute or chronic medical or psychiatric condition including recent (within the past year) or active suicidal ideation or behavior or laboratory abnormality that may increase the risk associated with study participation or investigational product administration or may interfere with the interpretation of study results and, in the judgment of the investigator, would make the participant inappropriate for entry into this study. Psychiatric adverse experiences have been reported in patients treated with modafinil with many, but not all, with prior psychiatric history. Participants with a history of psychosis, depression, or mania are excluded from this study.
* Use of prescription or nonprescription drugs and dietary and herbal supplements within 7 days or 5 half lives (whichever is longer) prior to the first dose of investigational product. As an exception, acetaminophen/paracetamol may be used at doses of ≤1 g/day. Limited use of nonprescription medications that are not believed to affect participant safety or the overall results of the study may be permitted on a case by case basis following approval by the sponsor.
* Previous administration with lorlatinib within 30 days (or as determined by the local requirement) or 5 half lives preceding the first dose of lorlatinib used in this study (whichever is longer).
* Previous treatment with lorlatinib
* A positive urine drug test, as confirmed by a single repeat.
* Screening supine blood pressure (BP) ≥130 mm Hg (systolic) or ≥80 mm Hg (diastolic), following at least 5 minutes of supine rest. If BP is ≥130 mm Hg (systolic) or ≥80 mm Hg (diastolic), the BP should be repeated 2 more times and the average of the 3 BP values should be used to determine the participant's eligibility.
* History of pancreatitis (elevated amylase or lipase) or hyperlipidemia.
* Screening supine 12 lead ECG demonstrating PR interval >200 msec, corrected QT (QTc) >450 msec or a QRS interval >120 msec.
* History of cardiac arrhythmia (excluding asymptomatic sinus arrhythmia with heart rate >50, and occasional asymptomatic premature atrial contraction and premature ventricular contractions), history of atrioventricular (AV) block, history of symptomatic bradycardia, history of QTc prolongation.
* Participants with ANY of the following abnormalities in clinical laboratory tests at screening: Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level > upper limit of normal (ULN); Total bilirubin level > ULN; participants with a history of Gilbert's syndrome may have direct bilirubin measured and would be eligible for this study provided the direct bilirubin level is ≤ ULN.
* History of alcohol abuse or binge drinking and/or any other illicit drug use or dependence within 6 months of Screening. Binge drinking is defined as a pattern of 5 (male) and 4 (female) or more alcoholic drinks in about 2 hours. As a general rule, alcohol intake should not exceed 14 units per week for males or 7 units per week for females (1 unit = 8 ounces (240 mL) beer, 1 ounce (30 mL) of 40% spirit or 3 ounces (90 mL) of wine).
* As modafinil is a controlled substance, participants with a history drug abuse will be excluded.
* Blood donation (excluding plasma donations) of approximately 1 pint (500 mL) or more within 60 days prior to dosing.
* History of sensitivity to lorlatinib or modafinil.
* Unwilling or unable to comply with the criteria in the Lifestyle Considerations section of this protocol.
* Male participants with partners currently pregnant; male participants able to father children who are unwilling or unable to use a highly effective method of contraception as outlined in this protocol for the duration of the study and for at least 97 days after the last dose of investigational product or longer based upon the compound's half life characteristics, and refrain from sperm donation for the duration of the study and for at least 97 days after the last dose of investigational product.
* Investigator site staff members directly involved in the conduct of the study and their family members, site staff members otherwise supervised by the investigator, or Pfizer employees, including their family members, directly involved in the conduct of the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2019-08-22 (Actual); Primary Completion 2019-12-09 (Actual); Study Completion 2019-12-09 (Actual)

PRIMARY OUTCOMES:
Number of Participants With Treatment Emergent Treatment-Related Adverse Events (AEs) | Baseline up to 28 days after last dose of modafinil or lorlatinib.
  Treatment-related AE was any untoward medical occurrence attributed to study drug in a participant who received study drug. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to Y days after last dose that were absent before treatment or that worsened relative to pretreatment state. Relatedness to Drug X was assessed by the investigator (Yes/No). Participants with multiple occurrences of an AE within a category were counted once within the category.
Number of Participants With Clinically Significant Change From Baseline in Laboratory Abnormalities | Baseline up to 28 days after last dose of modafinil or lorlatinib.
  Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Number of Participants With Clinically Significant Change From Baseline in Vital Signs | Baseline up to 28 days after last dose of modafinil or lorlatinib.
  Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.

SECONDARY OUTCOMES:
Area Under the Curve From Time Zero to Extrapolated Infinite Time (AUCinf) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  AUCinf = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-inf). It is obtained from AUC (0-t) plus AUC (t-inf).
Maximum Observed Plasma Concentration (Cmax) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Maximum observed plasma concentration.
Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Area under the plasma concentration time-curve from zero to the last measured concentration (AUClast).
Apparent Oral Clearance (CL/F) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Plasma Decay Half-Life (t1/2) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time to Reach Maximum Observed Plasma Concentration (Tmax) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Time to Reach Maximum Observed Plasma Concentration (Tmax)
Apparent Volume of Distribution (Vz/F) of lorlatinib | 0 (pre-dose), 0.5, 1, 1.5, 2, 4, 6, 12, 24, 36, 48, 60, 72, 96, and 120 hours post-dose in both Period 1 and Period 2.
  Volume of distribution is defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. Apparent volume of distribution after oral dose (Vz/F) is influenced by the fraction absorbed.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Be-bru, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- [Derived] Rodrigues AD, Wood LS, Vourvahis M, Rowland A. Leveraging Human Plasma-Derived Small Extracellular Vesicles as Liquid Biopsy to Study the Induction of Cytochrome P450 3A4 by Modafinil. Clin Pharmacol Ther. 2022 Feb;111(2):425-434. doi: 10.1002/cpt.2440. Epub 2021 Nov 2. PMID 34623637
- [Derived] Li J, Pithavala YK, Gong J, LaBadie RR, Mfopou JK, Chen J. The Effect of Modafinil on the Safety and Pharmacokinetics of Lorlatinib: A Phase I Study in Healthy Participants. Clin Pharmacokinet. 2021 Oct;60(10):1303-1312. doi: 10.1007/s40262-021-01026-w. Epub 2021 May 3. PMID 33937953
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7461026